CLINICAL TRIAL: NCT05082272
Title: Pulmoner Hipertansiyon gelişmiş Bronkopulmoner Displazili Pretermlerin Ekokardiyografik ve Biyokimyasal değerIendirilmesi
Brief Title: The Role of Transthoracic Echocardiography in Diagnosis of Pulmonary Hypertension of Infants With Bronchopulmonary Dysplasia
Status: Completed | Type: Observational
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, süleyman sunkak, Specialist (pediatric cardiolog), Kayseri City Hospital
Other Study IDs: 6196
Record Dates: First submitted 2021-10-06; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Hypertension; Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary dysplasia; Pulmonary hypertension; Echocardiography
MeSH Terms: conditions — Hypertension, Pulmonary; Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biomarkers like kallistatin, NT-ProBNP, gelsolin, homocysteine, cystatin C levels were measured.
  Serum was taken for Kallistatin, gelsolin and cystatin C Plasma was taken for NT-proBNP and homocysteine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Preterm neonates with bronchopulmonary dysplasia with pulmonary hypertension: Preterm neonates who continued need for respiratory support persisting at 36 weeks corrected postmenstrual age and diagnosed with pulmonary hypertension on echocardiographic examination
- Preterm neonates with bronchopulmonary dysplasia and without pulmonary hypertension: Preterm neonates who continued need for respiratory support persisting at 36 weeks corrected postmenstrual age and whose echocardiographic examination were normal
- Healty preterm neonates: preterm neonates with neither bronchopulmonary dysplasia nor pulmonary hypertension

SUMMARY:
Pulmonary hypertension may develop in premature newborn infants due to impaired lung development. The diagnosis of this disease can actually be made with interventional methods.

In this study, we evaluated the importance of echocardiographic examination and blood laboratory tests in diagnosing this disease.

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia diagnosis was done by the same neonatologist according to the criteria published by the American National Institutes of Health (NIH) in 2001.

Demographic data of patients like: birth weight, gender, gestational age; neonatal morbidity like: surfactant administration, PDA and its treatment, duration of mechanical ventilation, diuretic usage, intraventricular hemorrhage and its grade, necrotizing enterocolitis (NEC) and its severity, any surgical procedures and late-onset sepsis were recorded.

Moreover; maternal and perinatal risk factors like presence of chorioamnionitis, maternal hypertension and administration of antenatal steroids were also recorded.

Echocardiography:

Echocardiographic measurements were performed with a GE Vivid-7 pro equipped with a 3-7 MHz for 2-dimensional and color flow Doppler mapping by the same pediatric cardiologist.

Investigations were done in parasternal long, short axis, four chamber, five chamber views using M mode and Doppler wave. Two-dimensional measurements were done according to the guidelines of American Society of Echocardiography. M mode views were obtained in parasternal long axis by putting cursor between mitral valve and apical to tips of the MV leaflets. Ejection fraction and end diastolic or end systolic volumes were calculated using the Teicholtz (Teich) method. Estimated Pulmonary artery systolic pressure can be determined by using the modified Bernoulli equation: 4V2, where V is the maximum velocity of the tricuspid valve regurgitation jet, measured by continuous wave Doppler, added to the estimated right atrial pressure.

The echocardiography parameters showing pulmonary hypertension are tricuspid velocity, mean pulmonary artery pressure (PAP), pulmonary vascular resistance, pulmonary acceleration time, pulmonary velocity time integral, fraction of area changes of Right ventricle (RV), RV myocardial performance index (TEI). Severe pulmonary hypertension affects not only RV but also LV systolic functions. Therefore we measured Left Ventricle (LV) eccentricity index and LV TEI parameters in order to see whether they were affected in patients w BPD and PHT.

Pulmonary vascular resistance (PVR) can be measured using Tricuspid Velocity (m/s) and Velocity Time IntegralRVOT (cm) PVR (Wood units) = 10 × (TRV/VTIRVOT) + 0.16. Here, a TRV/VTIRVOT<0.2 corresponds approximately to a PVR of <2 Wood Units [8].

Left Ventricular Eccentricity index (EI), measured at end-systole and end-diastole, from the parasternal short axis 2D image at the mid-papillary muscle level. The formula (EI=D2/D1) was used where D1 is the ventricular diameter perpendicular to the interventricular septum bisecting D2: the diameter parallel to the interventricular septum [9].

RV systolic dysfunction occurs in PHT and shown by RV Fraction of Shortening (FS), tricuspid annular plane systolic excursion (TAPSE) and Inferior vena cava distensibility index.

Inferior vena cava distensibility index is calculated by measuring the Dmax and Dmin of IVC from the subcostal view, and IVCDI exceeding 18% has been reported to be predictive of fluid responsiveness in adults, and it is often extrapolated in children as well. IVCDI=Dmax-Dmin/Dmin [10].

First echocardiograms were performed at 36 to 38 weeks' post-menstrual age (PMA) for screening later repeated at 1, 3, 6 months after the first echocardiogram. Measurements were made during 3 consecutive cycles and mean values were used in statistical analysis.

Pulmonary hypertension diagnosis was done according to presence of at least one of the following criteria [11]: 1) the velocity of tricuspid valve regurgitation of ≥3 m/s in the absence of pulmonary stenosis or 2)estimated right ventricular systolic pressure (RVSP) greater than 40 mm Hg, or RVSP/systemic systolic blood pressure greater than 0.5, any 3) cardiac shunt with bidirectional or right-to-left flow, 4) flat or left-deviated interventricular septal configuration and right ventricular hypertrophy with chamber dilation.

Serum Biomarkers:

Serum biomarkers like kallistatin, NT-ProBNP, gelsolin, homocysteine, cystatin C levels were measured only in the beginning of the study and not repeated in the following controls.

1. Serum Kallistatin Levels Blood for kallistatin level was taken to the tubes centrifuged at 4000 rpm for 10 min at 4°C. The serum was kept at -80°C as frozen until required. Kallistatin levels were determined by ELISA (R&D Systems, Inc. Minneapolis, USA) as previously described [12].
2. Plasma NT-ProBNP Levels Five ml blood sample was drawn from both patient and control groups for N terminal pro Brain natriuretic peptide (NT-ProBNP). Blood samples were centrifuged at +4°C and 1500 rpm for 5 minutes. Plasma part of the upper phase was taken in to another tube for NT-ProBNP calculation. Samples were preserved at -80°C till the study date. Later on, they were studied with ELISA method using Biomedica N-terminal pro BNP commercial kits (NT- ProBNP enzyme immuno assay kit Biomedica, Bratislava, Slovakia) and Elecsys® 1010 aoutoanalyzer (Roche Diagnostics, Basel, Switzerland). Results were expresses as fmol/ml (1fmol/ml=16.1pg/ml).
3. Serum Gelsolin Levels:

   Venous blood samples of the healthy individuals and patients were drawn on admission. The blood samples were immediately placed in sterile etylene diamin tetra asetic acid test tubes and centrifuged at 2000-3000 rpm for 20 minutes at 4°C to collect plasma. Plasma was stored at -80°C until assayed. The concentration of gelsolin in plasma was analysed by enzyme-linked immunosorbent assay using commercial kits (Hangzhou Eastbiopharm Co., Ltd, Hangzhou, Zhejiang, China) in accordance with the manufacturer's instructions.
4. Plasma Homocysteine Levels:

   Plasma Homocysteine was measured using an auto-biochemical analyzer (AU5800, Beckman Coulter Company, U.S.A.) by the enzymatic method. This method uses the S-adenosyl homocysteine (SAH) hydrolase reaction principle, in which SAH is hydrolyzed by hydrolytic enzymes into adenosine and Homocysteine; adenosine is immediately hydrolyzed into ammonia and hypoxanthine, and nicotinamide adenine dinucleotide (NADH) is converted to NAD by ammonia and glutamic dehydrogenase. The concentration of Homocysteine in the sample is proportional to the NADH transformation rate. The detection reagents were provided by DiaSys Diagnosis System GmbH (Shanghai) Co., Ltd.
5. Serum Cystatin-C Levels:

Cystatin C levels were determined with an immune nephelometry method on an ProSpec analyzer (BN ProSpec, Siemens, Frimley, United Kingdom) using latex enhanced particles coated with anti-cystatin C antibodies. The reference values for young healthy persons range from 0.53 to 0.95 mg/l. The coefficient of variation was 1.8% within one run and 2.0% during reproducibility tests. Freezing and long-term storage up to 25 years has a small impact on stability of cystatin C [13].

The study was approved by the local research Ethics Committee. All the parents were informed written consent were taken from each of them about participating in the study.

Statistical analysis:

Data analysis was performed using IBM SPSS Statistics Standard Concurrent User V 25 (IBM Corp., Armonk, New York, USA). Continuous variables were expressed either as mean ± standard deviation or median 25th-75th percentiles. Distribution of numerical data is evaluated by Shapiro Wilk normality test Q -Q graphics. Categorical variables were expressed as counts, proportions, and percentages. A Kruskal-Wallis test was used to determine whether or not there is a statistically significant difference between the medians of three or more independent groups with non-parametric values. If statistical significance was detected (p<0.05) Post Hoc Analysis - Tukey test was performed for pairwise comparisons. For the repeated measures analysis of a dependent group; Friedman test was used.

ELIGIBILITY:
1. BPD patients with PHT

   Inclusion Criteria:
   * Born ≤ 28 postmenstrual weeks
   * Respiratory support persisting at 36 weeks corrected postmenstrual age.
   * Echocardiographic examination consistent with pulmonary hypertension
2. BPD patients without PHT

   Inclusion Criteria:
   * Born ≤ 28 postmenstrual weeks
   * Respiratory support persisting at 36 weeks corrected postmenstrual age.
   * Normal echocardiographic examination
3. Healty preterms

   * Born ≤ 28 postmenstrual weeks
   * Do not need respiratory support persisting at 36 weeks corrected postmenstrual age
   * Normal echocardiographic examination

Exclusion Criteria:

* Congenital heart disease (with the exception of patent ductus arteriosus or patent foramen ovale)
* Structural lung and airway malformations (including tracheobrochomalacia)
* Congenital diaphragmatic hernia
* Chromosome abnormality

Ages: 28 Days to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm newborns followed in the neonatal intensive care unit
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Echocardiographic examination | 1 month
  Echocardiographic examination is effective in diagnosing pulmonary hypertension in preterms with bronchopulmonary dysplasia and is consistent with the clinical findings of the patients.
Serum kallistatin level | 1 month
  Serum kallistatin level is effective in diagnosing pulmonary hypertension in preterms with bronchopulmonary dysplasia and is consistent with the clinical findings of the patients.